CLINICAL TRIAL: NCT03936361
Title: STATINS USE IN INTRACEREBRAL HEMORRHAGE PATIENTS
Brief Title: Statins In Intracerbral Hemorrhage
Acronym: SATURN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: NINDS Stroke Trials Network (StrokeNet) (Other); Canadian Stroke Consortium (CSC) (Other); University of Cincinnati (Other); Medical University of South Carolina (Other); Yale University (Other); MetroHealth Medical Center (Other); UH, Cleveland Medical Center (Unknown); Corewell Health West (Other); West Virginia University (Other); Columbia University (Other); Weill Medical College of Cornell University (Other); New York Presbyterian Brooklyn Methodist Hospital (Other); Buffalo General Medical Center (Unknown); State University of New York - Upstate Medical University (Other); St. Joseph's Regional Medical Center, New Jersey (Other); Tufts Medical Center (Other); Massachusetts General Hospital (Other); UMass Memorial Health (Other); Brigham and Women's Hospital (Other); Baystate Medical Center (Other); University of Vermont Medical Center (Other); Lahey Hospital & Medical Center (Other); Augusta University Medical Center (Unknown); Prisma Health-Upstate (Other); The Moses H. Cone Memorial Hospital (Other); University of Virginia (Other); George Washington University (Other); University of Maryland, Baltimore (Other); Mount Sinai Hospital, New York (Other); NYU Langone Medical Center - Tisch Hospital (Unknown); Montefiore Medical Center (Other); NYU Langone Hospital - Brooklyn (Unknown); Froedtert Hospital (Other); Central DuPage Hospital (Other); Rush University Medical Center (Other); Loyola University (Other); Stanford University (Other); Mercy San Juan Medical Center (Unknown); Oregon Health and Science University (Other); Kaiser Permanente (Other); University of Southern California (Other); Cedars-Sinai Medical Center (Other); University of New Mexico (Other); Long Beach Memorial Medical Center (Other); University of California, Irvine (Other); Arrowhead Regional Medical Center (Other); Huntington Memorial Hospital (Other); Scripps Health (Other); University of California, San Diego (Other); Ochsner Health System (Other); St. Joseph's Hospital and Medical Center, Phoenix (Other); Desert Care Network (Unknown); Eden Medical Center (Unknown); San Francisco General Hospital (Other); University of California, San Francisco (Other); University of Louisville (Other); Ohio State University (Other); University of Iowa (Other); Sanford Medical Center Fargo (Unknown); University of Nebraska (Other); Tampa General Hospital (Other); University of Florida (Other); Jackson Health System (Other); Mayo Clinic (Other); Baptist Medical Center Jacksonville (Unknown); Wayne State University (Other); University of Michigan (Other); Mercy Health Saint Mary Grand Rapids (Unknown); Metro Health, Michigan (Other); University of Kentucky (Other); McLaren Health Care (Other); Regions Hospital (Other); Allina Health System (Other); University of Kansas (Other); University of Minnesota (Other); St. Cloud Hospital (Unknown); Milton S. Hershey Medical Center (Other); Abington Memorial Hospital (Other); Temple University (Other); University of Pennsylvania (Other); Lehigh Valley Hospital (Other); York Hospital, York, PA (Other); Thomas Jefferson University (Other); University of Pittsburgh (Other); St. David's HealthCare (Other); Baylor College of Medicine (Other); Tulane Medical Center (Unknown); The University of Texas Health Science Center at San Antonio (Other); OU Medical Center (Unknown); University of Utah (Other); Swedish Medical Center (Other); St. Mary's Medical Center (Other); Banner University Medical Center (Other); Intermountain Medical Center (Other); Legacy Emanuel Medical Center (Unknown); Sacred Heart Medical Center Springfield (Unknown); Harborview Injury Prevention and Research Center (Other); University of Wisconsin, Madison (Other); Aurora BayCare Medical Center (Other); Wake Forest University Health Sciences (Other); University of Alabama at Birmingham (Other); University of South Alabama (Other); Carolinas Medical Center (Other); Barnes-Jewish Hospital (Other); St. Luke's Hospital, Kansas City, Missouri (Other); University of Arkansas (Other); OSF Healthcare System (Other); Cox Medical Center South (Unknown); North Shore University Hospital (Other); Rhode Island Hospital (Other); Hartford Hospital (Other); Staten Island University Hospital (Other); Johns Hopkins University (Other); University of North Carolina, Chapel Hill (Other); University of Alberta (Other); The Ottawa Hospital (Other); London Health Sciences Centre (Other); Hamilton General Hospital (Unknown); Hopital de l'Enfant-Jesus (Other); Montreal Neurological Institute and Hospital (Other); Foothills Medical Centre (Other); University Health Network, Toronto (Other); Health Sciences Centre, Winnipeg, Manitoba (Other); Thunder Bay Regional Health Sciences Centre (Other); Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre (Unknown); Fraser Health (Other); Hopital de Chicoutimi (Unknown); Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Magdy H Selim, MD, PhD, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018C000515
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; 3-hydroxy-3-methylglutaryl-coenzyme A

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at 1:1 ratio to either continue the same statin drug and dosage that they are taking at the time of ICH onset or to discontinue it for up to 24 months after ICH. No placebo will be prescribed for those randomized to discontinue statins.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Statin (Active Comparator): The same statin agent and dose that subjects were using at the time of ICH onset.
  Interventions: Drug: Statins
- No-statin (No Intervention): Subjects will discontinue the statin agent that they were taking at the time of ICH onset. No placebo will be prescribed for these subjects.

INTERVENTIONS:
Drug: Statins — Statin drugs (already prescribed) at ICH onset will be either continued or discontinued by the participants following qualifying ICH
  Other Names: HMG CoA
  Arms: Statin

SUMMARY:
The SATURN trial aims to determine whether continuation vs. discontinuation of statin drugs after spontaneous lobar intracerebral hemorrhage (ICH) is the best strategy; and whether the decision to continue/discontinue statins should be influenced by an individual's Apolipoprotein-E (APOE) genotype.

An MRI ancillary study (SATURN MRI), in a subset of SATURN participants , will evaluate the effects of continuation vs. discontinuation of statin drugs on hemorrhagic and ischemic MRI markers of cerebral small vessel disease, and whether the presence/burden of hemorrhagic markers (i.e. cerebral microbleeds and/or cortical superficial siderosis) on baseline MRI influences the risk of ICH recurrence on/off statin therapy.

DETAILED DESCRIPTION:
SATURN is a multi-center, pragmatic, prospective, randomized, open-label, and blinded end-point assessment (PROBE) clinical trial. A total of 1,456 patients presenting within 7 days of a spontaneous lobar ICH while taking statins will be randomized to one of two treatment strategies: discontinuation vs. continuation of statin therapy (using the same agent and dose that they were using at ICH onset). Participating subjects will undergo baseline testing for APOE genotype and will be followed for 24 months to assess for the occurrence of recurrent symptomatic ICH or major adverse cerebro-/cardio-vascular events (MACCE) during the follow-up period. A subset of SATURN participants will participate in the optional MRI study, where they will undergo a baseline MRI within 7 days of randomization into SATURN and a repeat MRI at the end of the follow-up period.

Recruitment will take place at ~ 140 sites coordinated through the NIH/NINDS StrokeNet and the Canadian Stroke Consortium.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years.
2. Spontaneous lobar ICH confirmed by CT or MRI scan
3. Patient was taking a statin drug at the onset of the qualifying/index ICH
4. Randomization can be carried out within 7 days of the onset of the qualifying ICH
5. Patient or legally authorized representative, after consultation with the statin prescriber, agrees to be randomized to statin continuation (restart) vs. discontinuation

Exclusion Criteria:

1. Suspected secondary cause for the qualifying ICH, such as an underlying vascular abnormality or tumor, trauma, venous infarction, or hemorrhagic transformation of an ischemic infarct.
2. History of recent myocardial infarction (attributed to coronary artery disease) or unstable angina within the previous 3 months
3. Diabetic patients with history of myocardial infarction or coronary revascularization
4. History of familial hypercholesterolemia
5. Patients receiving proprotein convertase subtilisin kexin 9 (PCSK9) inhibitors
6. Known diagnosis of severe dementia
7. Inability to obtain informed consent
8. Patients known or suspected of not being able to comply with the study protocol due to alcoholism, drug dependency, or other obvious reasons for noncompliance, such as unable to adhere to the protocol specified visits/assessments.
9. Life expectancy of less than 24 months due to co-morbid terminal conditions.
10. Pre-morbid mRS >3
11. ICH score >3 upon presentation.
12. Contraindications to continuation/resumption of statin therapy, such as significant elevations of serum creatinine kinase and/or liver transaminases, and rhabdomyolysis
13. Woman of childbearing potential
14. Concurrent participation in another research protocol for investigation of experimental therapy.
15. Indication that withdrawal of care will be implemented for the qualifying ICH.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1456 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent symptomatic ICH | within 24 months

SECONDARY OUTCOMES:
Major Adverse Cerebro- and Cardio-Vascular Events | Within 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchina S, Yeatts SD, Foster LD, Janis S, Shoamanesh A, Khatri P, Bernstein K, Perlmutter A, Stever C, Heistand EC, Broderick JP, Greenberg SM, Leira EC, Rosand J, Lioutas VA, Salman RAS, Tirschwell D, Marti-Fabregas J, Selim M. Rationale and Design of the Statin Use in Intracerebral Hemorrhage Patients (SATURN) Trial. Cerebrovasc Dis. 2025;54(2):270-277. doi: 10.1159/000538195. Epub 2024 Mar 16. PMID 38493765
- [Background] Marchina S, Foster LD, Yeatts SD, Khatri P, Bernstein K, Perlmutter A, Heistand EC, Smith EE, Sharma M, Broderick JP, Lioutas VA, Marti-Fabregas J, Selim M, Shoamanesh A. SATURN MRI: study protocol for the statin use in intracerebral hemorrhage patients MRI ancillary study. Trials. 2025 Aug 30;26(1):323. doi: 10.1186/s13063-025-09024-0. PMID 40886018
- [Background] Zhao W, Yeatts SD, Broderick JP, Selim MH, Adeoye OM, Durkalski-Mauldin VL, Meinzer CN, Martin RH, Dillon CR, Cassarly CN, Pauls KH, Elm JJ. Optimal Randomization Designs for Large Multicenter Clinical Trials: From the National Institutes of Health Stroke Trials Network Funded by National Institutes of Health/National Institute of Neurological Disorders and Stroke Experience. Stroke. 2023 Jul;54(7):1909-1919. doi: 10.1161/STROKEAHA.122.040743. Epub 2023 Apr 20. PMID 37078281
- [Derived] Szejko N, Kirsch E, Falcone GJ. Genetic determinants of LDL cholesterol and risk of intracerebral haemorrhage. Curr Opin Lipidol. 2021 Aug 1;32(4):244-248. doi: 10.1097/MOL.0000000000000761. PMID 34010223